CLINICAL TRIAL: NCT06066632
Title: Analysis of Calcium Score Values of Severe Aortic Stenosis in Patients With and Without Cardiac Amyloidosis (CAUSATIVE Study)
Brief Title: Analysis of Calcium Score of Severe Aortic Stenosis in Patients With and Without Cardiac Amyloidosis (CAUSATIVE Study)
Acronym: CAUSATIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Serenelli, Doctor, University Hospital of Ferrara
Other Study IDs: 72/2022/Oss/AOUFe
Record Dates: First submitted 2023-09-15; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Amyloidosis Cardiac; Aortic Stenosis, Severe
Keywords: Amyloidosis; Aortic stenosis; Calcium Score; Low-flow low-gradient
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Aortic Valve Stenosis; Amyloidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - "Dual Pathology": * Age >65 years
  * Severe aortic stenosis at echocardiographic examination
  * TAVI o SAVR planned or already undergone TAVI/SAVR
  * ECG-gated cardiac CT and echocardiographic examinations available before TAVI/SAVR
  * Cardiac uptake at bone tracer scintigraphy with a Perugini score of 2 or 3.
- Group 2- "Control Group": * Age >65 years
  * Severe aortic stenosis at echocardiographic examination
  * TAVI o SAVR planned or already undergone TAVI/SAVR
  * ECG-gated cardiac CT and echocardiographic examinations available before TAVI/SAVR
  * Patients with no cardiac uptake at scintigraphy with bone tracer.

SUMMARY:
The concomitant presence of cardiac amyloidosis (CA) in patients with aortic stenosis (AS) may challenge the estimation of stenosis degree. In patients with dual pathology (AS + CA) the most frequent AS hemodynamic profile is paradoxical low-flow, low-gradient AS.

In this setting, estimating stenosis degree with cardiac ultrasound may be challenging and aortic valve calcium score estimation by cardiac CT is a valuable exam.

Preliminary findings from small case series showed that patients with severe AS and CA presented less valvular calcium deposition compared to patients with severe AS alone. On this basis, confirmation of these findings would have a huge clinical impact on diagnosis, choice of treatment strategy and understanding of the pathophysiology of these patients.

The aim of the study is to study the correlation between valvular calcium score (assessed by EKG-gated CT) and effective orifice area (assessed through echocardiogram) according to cardiac amyloidosis presence (in the overall population and among hemodynamic phenotypes of cardiac amyloidosis).

As secondary endpoints the study will sought to assess TAVI/SAVR efficacy, procedural complications, in-hospital mortality, all-cause death and heart failure hospitalization at 1 year, according to absence or presence of CA.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is the most common valvular pathology in the elderly population, and there is an anticipated increase in prevalence and associated costs for treating this condition in the future. In a non-negligible percentage of cases (approximately 15%), another pathology is associated, namely cardiac amyloidosis, especially in the wild-type ATTR form. Patients with both pathologies (AS+ATTR) have a worse prognosis compared to those with AS alone. Based on the available data up to now, ATTR-associated amyloidotic cardiomyopathy does not appear to significantly influence the immediate outcome of TAVI or short-term outcomes. However, among patients with amyloidosis, there is an increased frequency of heart failure in subsequent follow-ups. The mechanism behind this dual pathology remains unclear. Epidemiological similarities (advanced age) alone do not explain the association. It is possible that there is a direct causal link between amyloidosis and aortic stenosis (amyloidosis as a co-cause or contributing factor to valvular stenosis), or that the elevated intramyocardial strain due to degenerative valvular stenosis promotes amyloidogenesis and myocardial infiltration. Understanding the extent of valvular calcifications in individual cases would provide better insights into the pathogenesis of this dual pathology. There are also diagnostic implications. Amyloidosis could potentially complicate the accurate classification of the severity of aortic pathology. For example, patients with AS+ATTR often exhibit a "low-flow low-gradient" paradoxical hemodynamic profile. In these cases, estimating the valve area with an echocardiogram is challenging, and evaluating the valvular calcium score through CT assumes an important diagnostic role. Preliminary studies suggest that, for the same degree of stenosis severity, there may be a lower quantity of calcium in the valves of patients with AS+ATTR compared to those with AS alone. Preliminary studies suggest that, for the same degree of stenosis severity, there may be a lower quantity of calcium in the valves of patients with AS+ATTR compared to those with AS alone. In a 1:1 propensity matching of over 300 patients (mostly without aortic stenosis), those with amyloidosis had lower aortic valvular calcium scores (p<0.01). In a small series of 13 cases with AS+ATTR, 12 had aortic valvular calcium scores below the severity cut-offs recommended by the guidelines. If confirmed, traditionally used calcium score cut-offs may be inadequate, with significant implications for treatment selection and therefore prognosis.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age ≥65 years old
* severe AS
* planned or performed TAVI/SAVR
* at least one red-flag suggestive of CA
* availability of EKG-gated CT
* availability of echocardiogram performed before TAVI/SAVR
* availability of bone scintigraphy performed within 1 year from CT

Exclusion Criteria:

• suboptimal acoustic window that may undermine the assessment of AS severity and phenotype profiling

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Group 1 "DUAL PATHOLOGY"
  * Age >65 years
  * Severe aortic stenosis at echocardiographic examination
  * TAVI o SAVR planned or already undergone TAVI/SAVR
  * ECG-gated cardiac CT and echocardiographic examinations available before TAVI/SAVR
  * Cardiac uptake at bone tracer scintigraphy with a Perugini score of 2 or 3.
  Group 2 "CONTROL GROUP"
  * Age >65 years
  * Severe aortic stenosis at echocardiographic examination
  * TAVI o SAVR planned or already undergone TAVI/SAVR
  * ECG-gated cardiac CT and echocardiographic examinations available before TAVI/SAVR
  * patients with no cardiac uptake at scintigraphy with bone tracer.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between valvular calcium score and effective orifice area. | Up to 12 months
  Correlation between valvular calcium score (assessed by EKG-gated CT) and effective orifice area (assessed through echocardiogram) according to cardiac amyloidosis presence (in the overall population and among hemodynamic phenotypes of cardiac amyloidosis).

SECONDARY OUTCOMES:
TAVI/SAVR efficacy | At time of post-procedural echocardiographic assessment (through study completion, an average of 1 month)
  Echocardiographic mean and maximal aortic gradient (mmHg) will be assessed.
TAVI/SAVR efficacy | At time of post-procedural echocardiographic assessment (through study completion, an average of 1 month)
  Echocardiographic effective orifice valvular area (EROA) will be assessed and reported in cm2.
Procedural Complications | At an average of 12 months
  Procedural complications will be assessed as per VARC definitions
In-hospital Mortality | At an average of 12 months
  In-hospital Mortality will be assessed from hospital records
All-cause Mortality and Heart Failure Hospitalization | At an average of 12 months
  The composite of all-cause Mortality and Heart Failure Hospitalization will be assessed through clinical follow-up, hospital records, and telephone follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Serenelli, Doctor, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available from the principal investigator on reasonable request.

REFERENCES:
- [Background] Hussan et al. Aortic Valve Calcium Score Cut-Offs Used To Identify Hemodynamically Severe Aortic Stenosis May Not Apply In Patients With Cardiac Amyloidosis. ACC.20 World Congress of Cardiology (https://www.jacc.org/doi/abs/10.1016/S0735-1097%2820%2932791-1)
- [Result] Hussain M, Hanna M, Griffin BP, Conic J, Patel J, Fava AM, Watson C, Phelan DM, Jellis C, Grimm RA, Rodriguez LL, Schoenhagen P, Hachamovitch R, Jaber WA, Cremer PC, Collier P. Aortic Valve Calcium in Patients With Transthyretin Cardiac Amyloidosis: A Propensity-Matched Analysis. Circ Cardiovasc Imaging. 2020 Oct;13(10):e011433. doi: 10.1161/CIRCIMAGING.120.011433. Epub 2020 Sep 23. No abstract available. PMID 32967445